CLINICAL TRIAL: NCT04219527
Title: Quantitative Assessment and Dual-target Intervention for Impinged and Frozen Shoulders: A Longitudinal Study of Dual-target Ultrasound Guided Corticosteroid Injection for Shoulder Impingement Syndrome
Brief Title: Dual-target Ultrasound Guided Corticosteroid Injection for Shoulder Impingement Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201910036RINC
Record Dates: First submitted 2019-12-27; First posted 2020-01-07 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2019-12

CONDITIONS: Shoulder Impingement
Keywords: Shoulder impingement; Subacromial bursa; Biceps tendon
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual-Target injection (Experimental): Corticosteroid injection into the subacromial bursa and biceps tendon
  Interventions: Procedure: Dual-target injection

INTERVENTIONS:
Procedure: Dual-target injection — Intervention procedure: corticosteroid injection into the subacromial bursa and biceps tendon
  Device for guidance: high-resolution ultrasound Drug: 40 mg triamcinolone acetonide (a kind of corticosteroid) + 3 mL of lidocaine (the medication will be mixed with 40 mg triamcinolone acetonide)

SUMMARY:
Subacromial injection is considered one of the best treatments for patients with subacromial impingement syndrome. The subacromial bursa is located between the deltoid muscle and the supraspinatus tendon. It facilitates the gliding of the humeral head through the undersurface of the acromion. If the bursa is thickened, the patient may experience pain when he/she tries to raise the arm. In patients with subacromial impingement due to a thickened subacromial bursa, the physician can precisely inject the medication into the bursa using ultrasound guidance. Use of ultrasound guidance has been proven to yield a better effect of pain relief than the technique using guidance. A previous study found that even using ultrasound guidance to deliver medication, there were still many patients suffering from initial treatment failure or recurrence after the first successful injection. Because the pathophysiological mechanism of subacromial impingement is complexed, the proximal biceps tendon may be involved but is often ignored. Recently, the investigators published a randomized controlled trial comparing the effect of dual-target injection (proximal biceps tendon and subacromial bursa) with the standard subacromial injection in patients with subacromial impingement syndrome, and found that the dual target approach was safe and had a longer effective duration than the standard subacromial injection. In this regard, the investigators will conduct a longitudinal follow-up study to examine the long-term effectiveness of the dual-target corticosteroid injection for subacromial impingement syndrome.

DETAILED DESCRIPTION:
Introduction:

Subacromial injection is considered one of the best treatments for patients with subacromial impingement syndrome. The subacromial bursa is located between the deltoid muscle and the supraspinatus tendon. It facilitates the gliding of the humeral head through the undersurface of the acromion. If the bursa is thickened, the patient may experience pain when he/she tries to raise the arm. In patients with subacromial impingement due to a thickened subacromial bursa, the physician can precisely inject the medication into the bursa using ultrasound guidance. Use of ultrasound guidance has been proven to yield a better effect of pain relief than the technique using guidance. A previous study found that even using ultrasound guidance to deliver medication, there were still many patients suffering from initial treatment failure or recurrence after the first successful injection. Because the pathophysiological mechanism of subacromial impingement is complexed, the proximal biceps tendon may be involved but is often ignored. Recently, the investigators published a randomized controlled trial comparing the effect of dual-target injection (proximal biceps tendon and subacromial bursa) with the standard subacromial injection in patients with subacromial impingement syndrome, and found that the dual target approach was safe and had a longer effective duration than the standard subacromial injection. In this regard, the investigators will conduct a longitudinal follow-up study to examine the long-term effectiveness of the dual-target corticosteroid injection for subacromial impingement syndrome.

Material and methods:

Participants: adult patients (>20 year old) with shoulder impingement syndrome Inclusion criteria: shoulder pain>3 weeks; no contraindication for local injection; Visual analogue scale of pain>4 The healthy volunteers are defined as no shoulder pain, and are only for the assessment of the inter-rater and intra-rater reliability of the ultrasound evaluation, without intervention

Participant number: 210 (150 with subacromial impingement, and 60 of healthy subjects) Exclusion criteria: systemic rheumatologic disease, Ankylosing spondylitis, malignancy, major trauma or recent injections on the affected shoulder

Study design:

The aims of this study is (1) set up the inter-rater and intra-rater reliability of the ultrasound evaluation in patients with subacromial impingement and healthy subjects (2) longitudinal follow up the therapeutic effect of dual-target injection to subacromial bursa and biceps tendon sheath only in patients with subacromial impingement

Detail of the intervention Single arm experiment: ultrasound guided injection into the subacromial bursa and biceps tendon sheath in patients with subacromial impingements, with 40 mg triamcinolone acetonide plus 3 mL of lidocaine

Outcome measurement:

physical examination(bicipital groove compression test, Speed's test, Yergason's test, empty can test, Neer's impingement test, Hawkins-Kennedy impingement test, painful arc test), range of motion as the baseline information. Visual analogue scale of pain, shoulder pain and disability index (SPADI), shoulder sonography (gray-scale/elastography)

Statistical analysis:

Continuous variables

1. Student's t test: fit assumption of normal distribution
2. Mann-Whitney test: does not fit the assumption of normal distribution

Categorical variables

(1) Chi-square test (2) Fisher exact test: sparse data

Multivariate analysis:

1. Linear regression
2. Logistic regression

Keywords: ultrasonography, corticosteroid, subacromial impingement syndrome, shoulder pain, longitudinal follow-up

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain>3 weeks; no contraindication for local injection; Visual analogue scale of pain>4

Exclusion Criteria:

* systemic rheumatologic disease, Ankylosing spondylitis, malignancy, major trauma or recent injections on the affected shoulder

The healthy volunteers are defined as no shoulder pain, and are only for the assessment of the inter-rater and intra-rater reliability of the ultrasound evaluation, without intervention.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in shoulder pain and disability index (SPADI) | Within 1 year after injection
  Shoulder pain and disability index (SPADI). The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability.

SECONDARY OUTCOMES:
Change in visual analogue scale of pain | Within 1 year after injection
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be' . The patient is asked to mark his pain level on the line between the two endpoints.
Doppler image of the rotator cuff tendons | Within 1 year after injection
  Doppler image of the rotator cuff tendons is to evaluate the vascularity, before and after treatment.
Elasticity (strain ratio) of the rotator cuff tendons | Within 1 year after injection
  Elasticity (strain ratio) is calculated for the target by selecting a region of interest (ROI) over the rotator interval and rotator cuff tendon, with a corresponding ROI of the adjacent reference tissue. The Using machine inherent software, the strain ratio value is displayed on a static image. The elasticity is measured before and after treatment.
Dynamic ultrasound evaluation | Within 1 year after injection
  The dynamic ultrasound evaluation is motion analysis regarding the related shoulder structures during shoulder abduction. The dynamic movement movie will be analyzed by software. The motion analysis is measured before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Vin Chang, Principal Investigator — National Taiwan University Hospital Bei-Hu Branch
Locations (1):
- National Taiwan University Hospital, Bei-Hu branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu WT, Lin CY, Shu YC, Chen LR, Ozcakar L, Chang KV. Predictive value of subacromial motion metrics for the effectiveness of ultrasound-guided dual-target injection: a longitudinal follow-up cohort trial. Insights Imaging. 2025 Jul 1;16(1):145. doi: 10.1186/s13244-025-01989-5. PMID 40593369